CLINICAL TRIAL: NCT06830915
Title: Evaluation of Current Practice of Antimicrobial Use and Clinical Outcome in the Management of Pneumonia Among Pediatric Patients Admitted to Jimma Medical Center, Southwest Ethiopia: A Prospective Observational Study
Status: Completed | Type: Observational
Sponsor: Bule Hora University (Other)
Collaborators: Jimma University (Other)
Responsible Party: Principal Investigator, Abduba Wariyo Guyo, Principal investigator, Bule Hora University
Other Study IDs: Ref. No. JUIRB016/21
Record Dates: First submitted 2025-02-12; First posted 2025-02-17 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Pneumonia; Bacterial
Keywords: Antimicrobial; use; Current; practice; Jimma; Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation only — No intervention made

SUMMARY:
A prospective observational study design was conducted on children admitted to the pediatric wards of Jimma Medical Center. The study was conducted from February 03, 2022, to June 03, 2022, and patients aged < 18 years and diagnosed with pneumonia were included. A chart review supplemented by a self-administered questionnaire was used to collect data. Descriptive statistics and binary logistic regressions were performed for data analyses.

DETAILED DESCRIPTION:
2.2 Study Design A hospital-based prospective observational study was conducted in children with pneumonia admitted to the pediatric ward of Jimma Medical Center.

2.3 Participant Eligibility and Inclusion All pediatric patients admitted to the pediatric ward of the Jimma Medical Center with a diagnosis of pneumonia during the study period were screened for eligibility criteria. Patients aged less than or equal to 18 years admitted to the pediatric wards of Jimma Medical Center with a suspected or proven pneumonia diagnosis by physician decision on duty during the study period and Patients whose parents gave assent were included in the study. Patients who died before they started antimicrobial, transferred to other facilities and patient lost follow-up were excluded.

2.4 Sample Size and Sampling Technique No sampling technique was applied; instead, all pediatric patients diagnosed with pneumonia that fulfilled illegibility criteria during the study period were recruited in the study. Accordingly, 146 patients were followed and completed data collected.

2.5 Data Collection Instrument and Quality Assurance The data collections instrument (data abstraction format and self-administered questionnaire) was developed by reviewing the literature on antimicrobial use, antimicrobial resistance, and antimicrobial stewardship program guidelines. Training was given for data collectors on the data collection procedure and research objectives. The principal investigator was regularly checking the consistency and completeness of the data and random checks were also being performed.

2.6 Data Processing and Analysis Data was compiled, cleared, coded, and verified for completeness and accuracy before being included in Epi Data Manager version 4.6.2. Double-entry verification was performed and the data was analyzed using statistical software, SPSS version 25.0. Descriptive statistics (mean, frequency, and cross tabulation) were used to describe practice of antimicrobial use. The bivariate logistic regression was performed for clinical outcome and variables with p-values less than 0.25 with outcomes (poor outcome or good outcome) were taken into account for further analysis. Then, the independent predictors were identified by multivariate logistic regression analysis. All statistical tests were detailed; a P value of less than or equal to 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged less than or equal to 18 years admitted to the pediatric wards of Jimma Medical Center with a suspected or proven pneumonia diagnosis by physician decision on duty during the study period and Patients whose parents gave assent were included in the study.

Exclusion Criteria:

* Patients who died before they started antimicrobial, transferred to other facilities and patient lost follow-up were excluded.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All pediatric patients admitted to the pediatric ward of the Jimma Medical Center with a diagnosis of pneumonia during the study period were screened for eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Antibiotics use pattern | February 03,2022 to June 03,2022
  Current practice of antimicrobial agents
Clinical outcome | February 03,2022 to June 03,2022
  Clinical treatment outcome(As poor vs good)

CONTACTS AND LOCATIONS:
Locations (1):
- Jimma University, Jimma, Oromiya, Ethiopia

IPD SHARING:
Plan to Share IPD: No